CLINICAL TRIAL: NCT00398827
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Dexmedetomidine for Sedation During Monitored Anesthesia Care
Brief Title: A Safety and Efficacy Study of Dexmedetomidine in Patients Requiring Sedation During Monitored Anesthesia Care (MAC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-005
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Anesthesia; Surgical Procedures, Elective
Keywords: American Society of Anesthesiologists (ASA); Observer's Assessment of Alertness Scale (OAA/S); Aldrete Scoring System; Surgery or procedure using monitored care anesthesia; Surgery or procedure at least 30 minutes in duration
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Dexmedetomidine 0.5 mcg/kg load (Experimental)
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 1 mcg/kg load (Experimental)
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: Dexmedetomidine 0.5 mcg/kg load; Dexmedetomidine 1 mcg/kg load
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of dexmedetomidine as compared to placebo when used for the sedation of subjects requiring monitored anesthesia care (MAC).

DETAILED DESCRIPTION:
Monitored anesthesia care (MAC) is a specific anesthesia service that involves an anesthesiologist administering sedatives and analgesics to a patient while monitoring his/her vital signs. MAC is often used to supplement local and regional anesthesia for non-intubated patients undergoing non-invasive procedures and minor surgery. The goal of MAC is to relieve anxiety by inducing a minimally depressed level of consciousness while the patient is able to continuously and independently maintain a patent airway and to respond appropriately to verbal commands.

Respiratory depression is the major concern with most of the medications (midazolam, fentanyl, propofol) currently used for MAC. There is clearly an unmet need for a sedative agent that can safely be used during MAC in both healthy and high risk populations with limited adverse side effects. A medication that can attenuate anxiety and the stress response associated with surgery and procedures without causing respiratory depression is highly desirable. A medication that reduces the total amount of opioids administered during a procedure could substantially reduce complications. Such a medication could be used either alone or in combination with other agents, thereby reducing the dose and side effects of the other agents.

Dexmedetomidine (DEX) has sympatholytic, sedative, analgesic, and anxiolytic effects that attenuate the catecholamine response to perioperative stress. DEX has not been associated with respiratory depression when used alone, despite sometimes deep levels of sedation.

An estimated 325 patients (260 DEX, 65 PBO) requiring MAC sedation for an elective surgery/procedure will be randomized at approximately 25 investigative sites.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age)
* American Society of Anesthesiologists (ASA) Physical Status I, II, III, or IV.
* If female, subject is non-lactating and is either:

  1. Not of childbearing potential, defined as post-menopausal for at least 1 year or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy or hysterectomy.
  2. Of childbearing potential but is not pregnant at time of baseline and is practicing one of the following methods of birth control: oral or parenteral contraceptives, double-barrier method, vasectomized partner, or abstinence from sexual intercourse.
* Subject requires monitored anesthesia care (MAC) in an operating room (OR) or procedure room with an anesthesiologist in attendance.
* Subject requires one of the following types of elective surgeries/procedures expected to take longer than 30 minutes:

  * Orthopedic
  * Ophthalmic
  * Plastic
  * Vascular stents
  * Breast biopsies
  * AV fistulas
  * Excision of lesion.
* Subject requires local anesthetic block.
* Subject (or subject's legally authorized representative) has voluntarily signed and dated the informed consent document approved by the Institutional Review Board.

Exclusion Criteria:

* Subject has received general anesthesia within 7 days prior to study entry, has received any experimental drug within 30 days prior to study drug administration, or has been previously enrolled in this study.
* Subject requires endotracheal intubation or laryngeal mask airway (LMA)
* Subject has central nervous system (CNS) disease with an anticipated potential for increased intracranial pressure, an uncontrolled seizure disorder, and/or known psychiatric illness that could confound a normal response to sedative treatment.
* Subject requires epidural or spinal anesthesia.
* Subject has received treatment with an alpha-2 agonist or antagonist within 14 days of the scheduled surgery/procedure.
* Subject for whom opiates, benzodiazepines, dexmedetomidine, or other alpha-2 agonists are contraindicated.
* Subject has received an intravenous (IV) opioid within one hour, or a by mouth (PO)/intramuscular (IM) opioid within 4 hours, of the start of study drug administration.
* Subject has acute unstable angina, acute myocardial infarction documented by laboratory findings in the past 6 weeks, heart rate <50 bpm, systolic blood pressure (SBP) <90 mmHg, or third-degree heart block unless patient has a pacemaker.
* Subject has known elevated serum glutamic pyruvic transaminase (SGPT/Alanine aminotransferase [ALT]) and/or serum glutamic oxaloacetic transaminase (SGOT/aspartate Aminotransferase [AST]) values of ≥2 times the upper limit of normal within the 2 months prior to screening, and/or a history of liver failure.
* Subject has any other condition or factor which, in the Investigator's opinion, might increase the risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2006-12; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Percent of patients not requiring midazolam for rescue sedation based on achieving and/or maintaining an Observer's Assessment of Alertness/Sedation Scale (OAA/S) score ≤4 | Prior to start of study drug, 15 minutes after start of study drug infusion, every 5 minutes thereafter throughout the study drug infusion and every 15 minutes while the subject is in the post anesthesia care unit.
  Observer's Assessment of Alertness/Sedation Scale (OAA/S) score ≤4 (Responsiveness: Lethargic response to name spoken in normal tone; Speech: Mild slowing or thickening; Facial Expression: Mild relaxation; Eyes: Glazed or mild ptosis [less than half the eye])

SECONDARY OUTCOMES:
Total amount (mg) of rescue midazolam required to achieve and/or maintain sedation (OAA/S score ≤4) | Prior to start of study drug, 15 minutes after start of study drug infusion, every 5 minutes thereafter throughout the study drug infusion and every 15 minutes while the subject is in the post anesthesia care unit.
Time from onset of study drug infusion to first dose of rescue midazolam | After the first 15 minutes of study drug infusion
  Subjects who are not adequately sedated (OAA/S is >4) may receive rescue MDZ (after attempting to achieve sedation via study drug titration).
Percentage of subjects who convert to alternative sedative and/or anesthetic therapy due to failure of treatment with study drug and rescue | Prior to start of study drug, 15 minutes after start of study drug infusion, every 5 minutes thereafter throughout the study drug infusion and every 15 minutes while the subject is in the post anesthesia care unit.
Time to recovery and readiness for discharge from Post-Anesthesia Care Unit (PACU) | Performed every 15 minutes while the subject is in the PACU until subject is discharged.
  Assessed by time from discontinuation of study drug to reach Aldrete score ≥9.
Total amount of fentanyl required for pain control | After the first 15 minutes of study drug infusion
Anesthesiologist assessment of ease of management | Approximately 24 hours
Anesthesiologist assessment of subject cooperation | Approximately 24 hours
Incidence of post-operative nausea and vomiting (PONV) in the PACU and during the 24 hour follow up | Approximately 24 hours
Overall Subject satisfaction and anxiety assessed 24 hours after study drug has been discontinued | 24 hours after study drug has been discontinued

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - University of Alabama, Birmingham, Alabama
  - Loma Linda Medical Center, Loma Linda, California
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami, Miami, Florida
  - South Miami Hospital, Miami, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Crossroads Research Inc., Owings Mills, Maryland
  - Chesapeake Research Group, Pasadena, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Missouri Health Care, Columbia, Missouri
  - NYU School of Medicine, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - VAMC, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dallas VA Medical Center, Dallas, Texas
  - Baylor Research Institute, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - University of Virginia, Charlottesville, Virginia
  - VA Medical Center, Milwaukee, Wisconsin